CLINICAL TRIAL: NCT00991419
Title: A Phase II, Open Label, Non-Randomized Study of [18F]AZD4694 to Compare PET Measurements of Fibrillar Amyloid Burden Obtained Using Difference Scanning Parameters, Reference Region Procedures and to Assess Test-retest Reliability in Patients With AD & HV
Brief Title: To Compare Positron Emission Tomography (PET) Measurements of Fibrillar Amyloid Burden
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: D2750N00006
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Alzheimer's Disease
Keywords: PET; Alzheimer's disease; diagnostic
MeSH Terms: conditions — Alzheimer Disease; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): [18F]4694
  Interventions: Drug: [18F]AZD4694

INTERVENTIONS:
Drug: [18F]AZD4694 — [18F]AZD4694 PET Ligand administered at Visit 1, 30 days following screening and at visit 4 for some of the participants.

SUMMARY:
The purpose of this study is to compare PET measurements of fibrillar amyloid burden using [18F]AZD4694.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, of any race or/ethnicity
* ECG, vital signs, and clinical laboratory values are within normal limits at enrollment or deemed not clinically significant by the physician

Exclusion Criteria:

* Significant recent (within 6 months) history of neurological (including stroke) or psychiatric disorder or substance abuse
* Participated in a PET study within the last 12 months
* Pregnancy or lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
PET Measurements | Day 1 and Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Reiman, MD, Principal Investigator — Banner Alzheimer's Institute
Locations (1):
- Research Site, Phoenix, Arizona, United States